CLINICAL TRIAL: NCT04617262
Title: Pilot Feasibility Study of Remote Problem Management Plus to Improve Well-being and Functioning of Adults Affected by COVID-
Brief Title: Pilot Feasibility Study of Remote Problem Management Plus for Adults Affected by COVID-19
Acronym: PM+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The New School (Other)
Collaborators: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-91-PM+
Record Dates: First submitted 2020-11-02; First posted 2020-11-05 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Depression; Anxiety Disorders; Psychological Distress
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote Problem Management Plus (Experimental): Five individual sessions of low-intensity psychological intervention
  Interventions: Behavioral: Remote Problem Management Plus

INTERVENTIONS:
Behavioral: Remote Problem Management Plus — Five sessions of low-intensity, trans-diagnostic psychological intervention including the teaching and practice of the following strategies: stress management, problem solving, behavioral activation, and strengthening social support

SUMMARY:
This is a pilot feasibility study of remotely delivered Problem Management Plus, a low-intensity psychological intervention, delivered in five sessions to adults affected by crisis. The current study will evaluate the feasibility and acceptability of the intervention when delivered remotely via Zoom to community members in New York City impacted by the COVID-19 pandemic. The investigator's goal is to use qualitative and quantitative approaches to inform procedures for a subsequent cluster randomized control trial of Problem Management Plus versus enhanced usual care. A mixed-methods design will be used to evaluate the feasibility, acceptability, perceived utility, and impact of the remotely delivered PM+ intervention, to determine recruitment and retention rates, to assess ethics and safety of trial procedures. Additionally, the study will evaluate the acceptability, feasibility and fidelity of the remote training and supervision of helpers trained to deliver the intervention.

DETAILED DESCRIPTION:
Problem Management Plus (PM+) is recommended as part of the World Health Organization Mental Health Gap Action Program for communities affected by adversity. It is a low-intensity, scalable manualized intervention that was designed according to a task-sharing model of care. PM+ has four core features that make the intervention suitable for populations exposed to adversities in low-resource settings. First, it is a brief intervention (five sessions); second, it can be delivered by paraprofessionals (trained, non-specialist workers, lay or peer providers under the supervision of a mental health professional), using the principle of task shifting/task sharing; third, it is designed as a trans-diagnostic intervention to address a range of client-identified emotional (e.g. depression, anxiety, traumatic stress, general stress) and practical problems; and, fourth, it is designed for communities affected by any kind of adversity (e.g. violence, disasters) in low-income countries. The intervention was originally developed for adults affected by humanitarian crises and tested in low-income countries. A number of randomized controlled trials in Kenya, Pakistan, Nepal, as well as the Netherlands have indicated that PM+ delivered by non-specialist helpers is effective in decreasing symptoms of psychological distress (including depression, anxiety and post-traumatic stress disorder symptoms) and improving functioning; however, empirical evidence of the feasibility and efficacy of the remote training and delivery of PM+ is limited.

In May 2020, the United Nations released a policy brief emphasizing inclusion of mental health and psychosocial support (MHPSS) in national response plans including scaling up access to remote support (UN, 2020). The brief was released in response to emerging concerns of the negative mental health and psychosocial impacts arising from the health and societal consequences of COVID-19. Extant population-based research is showing high rates of anxiety, depression, and general distress in the US, while at the same time MHPSS provision has been disrupted or halted due to social distancing measures. Remote delivery forms of PM+ may serve as an important mechanism to facilitate access to care during the ongoing pandemic and into the future. Furthermore, there is very limited research with PM+ in high-income countries where specialized mental health interventions are available, but where access for certain populations or during periods of public health crisis is limited due to systemic and practical barriers. Even in high income countries, only 22.4% of those with depression receive minimally adequate care; however, 64.9% of those with depression perceive a need for treatment. The treatment gap may be considerably higher among marginalized groups and economically disadvantaged communities. COVID-19 continues to bring on widespread mental health disparities, particularly among vulnerable and underserved communities that are disproportionately affected by COVID-19. Brief, low-intensity interventions designed to be implemented by non-specialists represent a promising and scalable approach to minimize this treatment gap in under-served US populations by partnering with community-based organizations (CBO) to train and supervise staff already involved in social and public health services. An important first step before investing resources in training and implementation with CBOs is to evaluate the feasibility, acceptability and effectiveness of remotely delivered PM+ with relevant community samples.

This is the first study to evaluate remotely delivered PM+ implemented by helpers whose training and supervision was conducted entirely online, as well as one of the first trials evaluating PM+ with community samples in the US. The aims of this pilot feasibility study are to a) assess interest from perspective beneficiaries by partnering with community-based organizations in New York City to recruit participants; b) to gather and evaluate information about the feasibility, acceptability and safety of the intervention, in particular when implemented via remote delivery; c) to identify whether the clinical and content adaptations that were made during the remote training, adaptation and conduct of initial practice cases are appropriate for the setting; and d) to assess possible problems of recruitment, delivery of the intervention and retention to ensure that procedures are adequate for a cluster randomized control trial. Additionally, the investigators will employ a single-arm, uncontrolled design in order to begin to examine the effectiveness and impact of remotely delivered PM+ among community members in New York City who are experiencing symptoms of common mental health problems. Lastly, trainees' knowledge and perceived self-efficacy in a) foundational helping skills based on common therapeutic factors and b) intervention-specific competencies will be evaluated pre-training, post-training and post-supervision.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Help- or treatment-seeking
* Access to a device for conducting sessions via Zoom (e.g., smartphone, tablet, laptop or personal computer)

Exclusion Criteria:

* Acute medical conditions or severe cognitive impairment (e.g., severe intellectual disability or dementia)
* Imminent suicide risk or expressed acute needs/protection risks (e.g., intimate partner violence risk)
* Presence of severe mental disorder (e.g., psychotic disorders)
* Hazardous substance use, substance dependency or substance use disorder (assessed using the Drug Abuse Screening Test (DAST-10) and Alcohol Use Disorders Identification Test (AUDIT-C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Psychological Outcomes Profile; Unabbreviated scale title "Psychological Outcomes Profile" | 1 week post-intervention
  4-item measure of personalized distress and client-generated problems, function and wellbeing; minimum value = 0, maximum value = 20; higher scores mean greater distress
Patient Health Questionnaire; Unabbreviated scale title "Patient Health Questionnaire" | 1 week post-intervention
  9-item measure of depression symptoms; minimum value = 0, maximum value = 27; higher scores mean more severe depression symptoms
Generalized Anxiety Disorder Scale; Unabbreviated scale title "Generalized Anxiety Disorder 7-item Scale" | 1 week post-intervention
  7-item measure of anxiety symptoms; minimum value = 0 and maximum value = 21; higher scores mean more severe anxiety symptoms

SECONDARY OUTCOMES:
World Health Organization Disability Assessment Scale 2.0; Unabbreviated scale title "World Health Organization Disability Assessment Scale 2.0" | 1 week post-intervention
  12-item measure of ability to engage in daily activities and functioning; minimum value = 0, maximum value = 48; higher scores mean worse disability outcomes
World Health Organization Quality of Life Questionnaire-BREF; Unabbreviated scale title "World Health Organization Quality of Life Questionnaire-BREF" | 1 week post-intervention
  26-item quality of life assessment of physical health, psychological health, social, relationships and environment; minimum value = 26 and maximum value = 130; higher scores mean better quality of life
EuroQoL 5-dimension 5-level; Unabbreviated scale title "EuroQoL 5-dimension 5-level" | 1 week post-intervention
  5-item assessment of dimensions of health status: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; minimum= 5, maximum = 25; higher score mean worse health outcomes
Pittsburgh Sleep Quality Index; Unabbreviated scale title "Pittsburgh Sleep Quality Index" | 1 week post-intervention
  19-item measure of sleep quality and disturbance; 19 items combined to form 7 "component" scores, each of which has a range of 0-3 points, 7 component scores are added to yield one global global score; minimum value = 0 and maximum value = 21; higher score means greater difficulty sleeping
Somatic Symptom Scale-8; Unabbreviated scale title "Somatic Symptom Scale-8" | 1 week post-intervention
  8-item assessment of the presence and severity of common somatic symptoms; minimum value = 0, maximum value = 32; higher score means more severe somatic symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Adam Brown, PhD, Principal Investigator — The New School; Brandon Kohrt, MD, PhD, Study Director — George Washington University
Locations (1):
- The New School, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data will be available through National Institute of Mental Health Data Archive after publication of primary results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Materials, de-identified patient data and results will be shared after publication of primary results, anticipated May 20, 2024.
Access Criteria: Contact investigators.

REFERENCES:
- [Background] Bryant RA, Schafer A, Dawson KS, Anjuri D, Mulili C, Ndogoni L, Koyiet P, Sijbrandij M, Ulate J, Harper Shehadeh M, Hadzi-Pavlovic D, van Ommeren M. Effectiveness of a brief behavioural intervention on psychological distress among women with a history of gender-based violence in urban Kenya: A randomised clinical trial. PLoS Med. 2017 Aug 15;14(8):e1002371. doi: 10.1371/journal.pmed.1002371. eCollection 2017 Aug. PMID 28809935
- [Background] Dawson KS, Schafer A, Anjuri D, Ndogoni L, Musyoki C, Sijbrandij M, van Ommeren M, Bryant RA. Feasibility trial of a scalable psychological intervention for women affected by urban adversity and gender-based violence in Nairobi. BMC Psychiatry. 2016 Nov 18;16(1):410. doi: 10.1186/s12888-016-1117-x. PMID 27863515
- [Background] Rahman A, Riaz N, Dawson KS, Usman Hamdani S, Chiumento A, Sijbrandij M, Minhas F, Bryant RA, Saeed K, van Ommeren M, Farooq S. Problem Management Plus (PM+): pilot trial of a WHO transdiagnostic psychological intervention in conflict-affected Pakistan. World Psychiatry. 2016 Jun;15(2):182-3. doi: 10.1002/wps.20312. No abstract available. PMID 27265713
- [Background] Dawson KS, Bryant RA, Harper M, Kuowei Tay A, Rahman A, Schafer A, van Ommeren M. Problem Management Plus (PM+): a WHO transdiagnostic psychological intervention for common mental health problems. World Psychiatry. 2015 Oct;14(3):354-7. doi: 10.1002/wps.20255. No abstract available. PMID 26407793